CLINICAL TRIAL: NCT04391036
Title: A Randomized Double-Blind Cross-Over Study of Self-Insertion of Two Formulations of a Placebo Vaginal Film
Brief Title: Randomized Cross-Over Study of Self-Insertion of Two Placebo Vaginal Film Formulations
Acronym: FAME103B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Katherine Bunge (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Katherine Bunge, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: STUDY20040030; 1U19AI120249 (NIH)
Record Dates: First submitted 2020-05-12; First posted 2020-05-18 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Safety; Acceptability
Keywords: Vagina; Film; Extended Release

STUDY DESIGN:
Intervention Model Description: Each participant will self-insert one low level Eudragit® and one high level Eudragit® formulation film. The sequence of insertion will be randomized in a 1:1 ratio.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participants, clinicians, and assessors of the study outcomes will be blinded to Eudragit® content of the film.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- High Eudragit® Film, then Low Eudragit® Film (Experimental): High (12.8%) Eudragit® content vaginal film, then low (6.4%) Eudragit® content vaginal film
  Interventions: Device: High Eudragit® Content Vaginal Film; Device: Low Eudragit® Content Vaginal Film
- Low Eudragit® Film, then High Eudragit® Film (Experimental): Low (6.4%) Eudragit® content vaginal film, then high (12.8%) Eudragit® content vaginal film
  Interventions: Device: High Eudragit® Content Vaginal Film; Device: Low Eudragit® Content Vaginal Film

INTERVENTIONS:
Device: High Eudragit® Content Vaginal Film — High (12.8%) Eudragit® Content Vaginal Film
Device: Low Eudragit® Content Vaginal Film — Low (6.4%) Eudragit® Content Vaginal Film

SUMMARY:
This is a double-blinded crossover study to evaluate whether Eudragit® content impacts the ability to self-insert placebo vaginal films. Thirty women will self-insert one high and and one low Eudragit® content film. The insertion order will be randomized in a 1:1 ratio. After inserting each film, participants will complete a survey reporting their perceptions and experience. The primary endpoint is successful insertion defined as all of the film inside the vagina upon visual assessment by a study clinician. Secondary outcomes include preference for the low level or high level Eudragit® formulation film with respect to insertion and participants' description of identified challenges.

DETAILED DESCRIPTION:
This is a double-blinded crossover study to evaluate whether ammonio methacrylate copolymer dispersion type B (Eudragit®) content impacts the ability to self-insert placebo vaginal films. Eudragit® is a commonly used pharmaceutical excipient, present in several FDA approved products. This hydrophobic excipient is used in vaginal film formulations to increase disintegration time and impart extended drug release property. The presence of Eudragit and its concentration level affects film disintegration and spreadability in the vaginal environment, and are likely to affect tactile properties. Consequently, these attributes may impact ease of film administration, acceptability, and user preferences for specific film type.

Thirty pre-menopausal women, 18 - 45 years of age, will self-insert one high and and one low Eudragit® content film. High and low Eudragit films correspond to 12.8% and 6.4% of Eudragit® added during the formulation blending stage. The insertion order will be randomized in a 1:1 ratio. Within 10 minutes of the insertion, clinical staff will perform a speculum exam to assess the location of the film and remove the residual film. After inserting each film, participants will complete a survey reporting their perceptions and experience. The primary endpoint is successful insertion defined as all of the film inside the vagina upon visual assessment by a study clinician. Secondary outcomes include preference for the low level or high level Eudragit® formulation film with respect to insertion and participants' description of identified challenges.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-45
* Intact uterus by participant report
* Agrees to abstain from inserting anything into the vagina for 24 hours prior to the study visit

Exclusion Criteria:

* Menopausal (as defined as amenorrhea for one year or more without an alternative etiology)
* Hysterectomy (including total and supracervical)
* Currently pregnant or pregnancy within 90 days of enrollment
* Lactating
* Symptoms of a urogenital infection including vaginal discharge, pain, odor, or itching
* Menses at the time of enrollment
* Known allergy or hypersensitivity to any of the components of the placebo film
* Any condition that, in the opinion of the Investigator, would preclude provision of consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Hillier, PhD, Principal Investigator — University of Pittsburgh; Katherine Bunge, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Magee Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Visness CM, Ulin P, Pfannenschmidt S, Zekeng L. Views of Cameroonian sex workers on a woman-controlled method of contraception and disease protection. Int J STD AIDS. 1998 Nov;9(11):695-9. doi: 10.1258/0956462981921224. PMID 9863584
- [Background] Nel AM, Mitchnick LB, Risha P, Muungo LT, Norick PM. Acceptability of vaginal film, soft-gel capsule, and tablet as potential microbicide delivery methods among African women. J Womens Health (Larchmt). 2011 Aug;20(8):1207-14. doi: 10.1089/jwh.2010.2476. Epub 2011 Jul 20. PMID 21774672
- [Background] Raymond E, Alvarado G, Ledesma L, Diaz S, Bassol S, Morales E, Fernandez V, Carlos G. Acceptability of two spermicides in five countries. Contraception. 1999 Jul;60(1):45-50. doi: 10.1016/s0010-7824(99)00060-8. PMID 10549452
- See also: UNAIDS Women and Girls and HIV. — https://www.unaids.org/sites/default/files/media_asset/women_girls_hiv_en.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Eudragit® Film, Then Low Eudragit® Film | Low Eudragit® Film, Then High Eudragit® Film
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Eudragit® Film, Then Low Eudragit® Film | Low Eudragit® Film, Then High Eudragit® Film | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (8.6) | 28.1 (5.3) | 29.8 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 15 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 8 | 8 | 16
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.3 (10.2) | 28.2 (5.6) | 29.7 (8.2)
Sexually Active [Count of Participants; unit: Participants] | 9 | 14 | 23
Prior participation in vaginal film studies [Count of Participants; unit: Participants] | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Successfully Insert Vaginal Film
Description: Number of participants that successfully insert each vaginal film defined as the film location being completely inside the vagina upon visual assessment by a clinician
Time Frame: Approximately 30 minutes
Population: All participants who attempted insertion of both vaginal film products which included the entire cohort of 30 enrolled participants.
Measure: Count of Participants; unit: Participants
Groups:
- High Eudragit® Film: High Eudragit® Content Vaginal Film: High (12.8%) Eudragit® Content Vaginal Film
- Low Eudragit® Film: Low Eudragit® Content Vaginal Film: Low (6.4%) Eudragit® Content Vaginal Film
Arm/Group | High Eudragit® Film | Low Eudragit® Film
Number analyzed (Participants) | 30 | 30
Participants
  Successful Insertion | 8 | 8
  Unsuccessful insertion | 22 | 22
Statistical Analysis 1: Comparison: High Eudragit® Film vs Low Eudragit® Film; This was a paired analysis comparing successful insertion of the high and low Eudragit® Films. The McNemar's test statistic is based on the discordant pairs (number of participants with high successful, low unsuccessful versus low successful, high unsuccessful); Test type: Superiority; p > .99, McNemar

2. Secondary Outcome: Number of Participants That Report Self-Insertion of Vaginal Film Was Easy
Description: Participants that report that self-insertion of the placebo vaginal film was not difficult at all as assessed on a Likert scale from 1 (not difficult at all) to 4 (very difficult)
Time Frame: Approximately 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | High Eudragit® Film | Low Eudragit® Film
Number analyzed (Participants) | 30 | 30
Participants
  Not Difficult To Insert | 11 | 8
  At Least Some Difficulty Inserting Film | 19 | 22
Statistical Analysis 1: Comparison: High Eudragit® Film vs Low Eudragit® Film; Test type: Superiority; p = .45, McNemar — This was a paired analysis comparing difficulty of insertion of the high and low Eudragit® Films. The McNemar's test is based on discordant pairs (high was not difficult, low was difficult versus low was not difficult, high was difficult)

3. Secondary Outcome: Number of Participants That Prefer the High Over the Low Eudragit® Content Vaginal Film
Description: Number of participants that report that they would prefer to use the high Eudragit® content vaginal film over the low Eudragit® content vaginal film. This outcome was analyzed by order of film product use (high then low vs low then high) as this may influence product preference.
Time Frame: Approximately 1 hour
Population: All participants that attempted insertion of both vaginal film products; this included the entire cohort of 30 enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | High Eudragit® Film, Then Low Eudragit® Film | Low Eudragit® Film, Then High Eudragit® Film
Number analyzed (Participants) | 15 | 15
Participants
  Preferred High Eudragit® Film | 5 | 9
  Preferred Low Eudragit® Film | 5 | 2
  No Preference | 5 | 4
Statistical Analysis 1: Comparison: High Eudragit® Film, Then Low Eudragit® Film vs Low Eudragit® Film, Then High Eudragit® Film; Test type: Superiority; p = .26, Fisher Exact; This was an overall Fisher's exact test so the analysis applies to all categories

ADVERSE EVENTS:
Time Frame: 1 week
Description: The arms were combined since participants used both films within a single visit which lasted 60-90 minutes. Within 10 minutes after the first film insertion, a speculum exam was performed to assess location of the film, then all film was removed. The participant then inserted the second film, and the aforementioned procedure was repeated. Thus, it was not possible to determine which film any adverse events would be attributable to. No adverse events were observed or reported during this study.
Arm/Group | High Eudragit® Film, Then Low Eudragit® Film | Low Eudragit® Film, Then High Eudragit® Film
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT04391036/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT04391036/ICF_001.pdf